CLINICAL TRIAL: NCT05650177
Title: Investigating Effects of Mindfulness Training on DMN Connectivity and Dynamics
Brief Title: Effects of Mindfulness on Brain Functioning in Depressed Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Surrey (Other)
Collaborators: Surrey and Borders Partnership NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: USurrey
Record Dates: First submitted 2022-11-30; First posted 2022-12-14 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: Persistent Depressive Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Receiving intervention. (Experimental): Patients with persistent depression who are receiving the intervention.
  Interventions: Behavioral: blended Mindfulness-Based Intervention (bMBI)

INTERVENTIONS:
Behavioral: blended Mindfulness-Based Intervention (bMBI) — The blended Mindfulness-Based Intervention (bMBI) is a 24-week online course 'blended' with therapist support via video link. The entire course is completed online and requires no in person contact. The bMBI follows the general structure of Mindfulness-Based Cognitive Therapy (MBCT) with an added emphasis on the cultivation of self-compassion. The bMBI comprises of 9-themed sessions spread out over the 24-weeks. Each session involves: video instructions, written information, psycho-educational exercises, and guided meditation practices. Participants meditate for 30-minutes each day. Additional homework involves short daily activities designed to incorporate mindfulness into daily life and keeping a journal about experiences within and around the practices and exercises. The therapist sessions are every two weeks and last for 45-minutes and help participants overcome any problems they experience.

SUMMARY:
Depression is a common disorder that often takes a recurrent or chronic course. Recent research has indicated that such courses are associated with significant changes in brain functioning including changes in strength of functional connectivity between regions of the default mode network, a large-scale brain network involved in spontaneous thinking and rumination, and the ability to suppress this network.

Training in mindfulness has been found to be an effective treatment for patients with recurrent and chronic courses of depression and there is evidence for beneficial effects on brain structure and functioning. However, it remains unclear whether and in how far the training may serve to reverse brain changes in recurrent and chronic courses of depression. The aim of this research is to test the effects of sustained training in mindfulness meditation on default mode network connectivity and suppression in patients suffering from recurrent or chronic depression.

The investigators will invite currently depressed patients with a recurrent or chronic course of the disorder (N = 36) to take part in a 6-month mindfulness intervention and investigate changes in default-mode network connectivity and suppression over repeated assessments. Building on our previous research, the intervention will use a blended format that combines an online app offering psychoeducational materials and meditation guidance with brief individual therapy sessions delivered via videoconference. Eligible participants will be asked to complete questionnaires and take part in brain scans before the start of the treatment, 3 months after the start of the treatment and after the end of treatment.

DETAILED DESCRIPTION:
Background and rationale

Major Depression is one of the leading contributors to the burden of disease world-wide. While there are established treatments, a considerable proportion of patients do not respond sufficiently. About a third of people who suffer from depression develop an increasingly chronic and recurrent course that is accompanied by progressive changes in brain structure and functioning. These changes act to prevent recovery and play an important role in conferring an increased risk for associated physical and neurodegenerative disorders.

Training in mindfulness helps patients recognize and disengage from the maladaptive and habitual patterns of thinking that maintain the disorder and has been shown to have promising effects in the treatment of such persistent courses. Mindfulness-Based Cognitive Therapy (MBCT), a standard MBI consisting of eight weekly sessions, is now a recommended treatment for the prevention of relapse in highly recurrent courses of depression.

However, recent research indicates that beneficial effects are contingent on sustained practice and utilization of mindfulness skills beyond the actual intervention periods. There is now an increasing awareness of the need to support patients in establishing a sustained practice of mindfulness. Yet despite the fact that this need is now widely acknowledged, there are currently no established approaches to support patients in sustained practice and it remains unclear in how far, and at what levels, sustained practice may lead to visible changes in underlying neurobiological vulnerabilities. While standard MBIs have been shown to have significant beneficial effects in patients with persistent forms of depression, there is still a considerable proportion of patients who do not respond sufficiently - current trials suggest a response rate of about 50%. Few studies have investigated reversibility of neurobiological vulnerabilities in depression. However, research in healthy meditators suggests that sustained practice in mindfulness may have promising potential for this purpose. Establishing approaches to support patients in sustained practice and understanding its effects on neurobiological vulnerabilities therefore represents an important step in improving MBIs for this group.

Previous research has indicated that the psychological maintenance mechanisms that hold persistent forms of depression in place are associated with significant changes in the connectivity and dynamics of the DMN, a large distributed network of interacting brain regions that serves to imbue present moment experience with memory content and becomes active when people engage in mind wandering and other forms of task-unrelated thinking such as rumination. Research in patients with depression has shown that depression is characterised by significant deficits in suppressing DMN activity during performance of common working memory and other executive tasks. Furthermore, there is now considerable evidence for aberrations in connectivity within and from this network to other regions of the brain that are relevant in the regulation of attention and emotions.

This study is the second stage of the project. In the first stage, the investigators tested the feasibility and acceptability of a blended Mindfulness-Based Intervention (bMBI) over a period of 3-months. The bMBI is an online course 'blended' with therapist support via video link. The online course comprises of 9 themed sessions each involving: video instructions, written information, exercises, and practices. The therapist sessions are biweekly and help participants overcome any problems they experience. In this stage, the investigators will investigate the effects of engaging in the bMBI over an extended period of 6-months on brain functioning using brain imaging techniques. The investigators will specifically look at the effects of the intervention on DMN suppression and connectivity in a sample of patients suffering from persistent depression.

ELIGIBILITY:
Inclusion Criteria:

1. A current diagnosis of Major Depression as assessed by SAGE-SR (Series of Assessments to Guide Evaluation Self Report (Brodey et al., 2018).
2. A chronic or recurrent lifetime history of depression, with either chronic persistence of symptoms or a history of at least three previous episodes of depression, two of which needed to have occurred during the last two years.
3. Self-reported severity of current symptoms on a clinical level as indicated by a PHQ-9 score of 10 or more.
4. Age 18 to 65 thus excluding cases of late life depression given that such cases might differ in aetiology.
5. Fluency in spoken and written English.
6. Have individual access to a computer or mobile device with internet connection and video link.
7. Fully committed to the intervention and assessments as assessed by the Participation Form.

Exclusion Criteria:

1. History of schizophrenia, schizoaffective disorder, bipolar disorder, current abuse of alcohol or other substances, organic mental disorder, pervasive developmental delay, primary diagnosis of obsessive-compulsive disorder or eating disorder, or regular non-suicidal self-injury.
2. Current treatment with CBT more than once a month.
3. Regular meditation practice (meditating more than once per week).
4. Inability to complete research assessments through difficulty with English, visual impairment, or cognitive difficulties.
5. We will allow patients who are currently taking antidepressants into the study provided that their medication has not been changed during the last four weeks before entry into the study.
6. People with heart pacemakers and clips or other metal items, which have been implanted into the body by a surgeon. This is because they would not safe in the brain scanner.
7. Suffer from claustrophobia.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2022-06-06 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Changes in activity within the brain's 'default mode network'. | 0 months, 3 months, and 6 months.
  The primary outcome measure is changes in activity within the brain's 'default mode network', measured during a working memory task. The default mode network (DMN) refers to an interconnected group of brain structures (including medial prefrontal cortex, posterior cingulate cortex, and the inferior parietal lobule) that is more active when we are not involved in any specific mental exercise, e.g. just daydreaming, recalling memories or thinking about the future. Research has found links between activity in the DMN and mental disorders including depression and anxiety, while mindfulness practise has been shown to influence DMN activity.

SECONDARY OUTCOMES:
Patient Health Questionnaire-9 (PHQ-9) | 0 months, 3 months, and 6 months.
  Reductions in depression symptomatology as assessed using the Patient Health Questionnaire-9 (PHQ-9).
Experiences Questionnaire (EQ) | 0 months, 3 months, and 6 months.
  Ability to decenter as assessed by self-report on the Experiences Questionnaire (EQ). The ability to decenter from thoughts and feelings (to see them as events that arise in the mind rather than being involved in them) is a key mechanism for which mindfulness has been found to be effective for mental health disorders.
Five-Facet Mindfulness Questionnaire (FFMQ-15) | 0 months, 3 months, and 6 months.
  Levels of mindfulness in daily life as assessed using the Five-Facet Mindfulness Questionnaire (FFMQ-15).
Amsterdam Resting-State Questionnaire 2.0 (ARSQ 2.0) | 0 months, 3 months, and 6 months.
  Mind wandering and spontaneous thoughts as assessed by the Amsterdam Resting-State Questionnaire 2.0 (ARSQ 2.0).
Generalised Anxiety Disorder Assessment (GAD-7) | 0 months, 3 months, and 6 months.
  Symptoms of anxiety as assessed using the Generalised Anxiety Disorder Assessment (GAD-7).
Perceived Stress Scale (PSS) | 0 months, 3 months, and 6 months.
  Subjective levels of stress as assessed using the Perceived Stress Scale (PSS).
Warwick-Edinburgh Mental Wellbeing Scale (WEMWBS) | 0 months, 3 months, and 6 months.
  Mental wellbeing as assessed using the Warwick-Edinburgh Mental Wellbeing Scale (WEMWBS).

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan D Hamilton, Principal Investigator — University of Surrey
Locations (1):
- University of Surrey, Guildford, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: No